CLINICAL TRIAL: NCT03259945
Title: Retrospective Observational Study of Patients With a Sutureless Aortic Valve Implanted in the Cardiovascular and Thoracic Surgery Department of Dijon CHU
Acronym: ORVAS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BOUCHOT 2017
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Patients With a Sutureless Aortic Valve
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — demographic and clinical data
Other: Review of ECGs — nature and frequency of proven conduction disorders

SUMMARY:
The incidence of aortic valve disease is increasing steadily because of the ageing of the population. At a certain stage, replacement of the aortic valve improves symptoms and thus the quality of life of patients.

Surgical aortic valve replacement is the " gold standard ". The procedure involves stopping the heart and setting up cardiopulmonary bypass (CPB) to ensure the oxygenation of tissues.

The reference technique consists in suturing a prosthetic valve to the aortic annulus so as to restore normal function. This technique has very good results in the long term. The elective approach is sternotomy, which has certain drawbacks: post-operative pain, risk of infection, psychological trauma of a major incision. In recent years an alternative approach, right minithoracotomy, has been proposed. The drawback to this approach is that it increases aortic cross-clamp time and CPB time.

More recently, new prosthetic valves, so-called "sutureless" or "rapid deployment" valves have become available. The main advantage of these valves is that they are easy to implant, as they do not require or need just a few sutures. As a result heart-arrest time is shorter, post-operative inflammatory syndrome is less frequent and transfusion needs are reduced.

However, these valves have a metallic stent to fix the valve in place by pressing against the aortic annulus, which may give rise to intra-cardiac conduction disorders. Yet, very few studies have been conducted on this subject.

The investigators wish to evaluate these conduction disorders in a cohort of patients operated on in this Department with this sutureless or rapid deployment valve technique.

ELIGIBILITY:
Inclusion Criteria:

All patients who underwent implantation of a Suturless valve since 2015 (Intuity Elite Edwards or Perceval S Liva Nova)

Exclusion Criteria:

* patients with a pacemaker
* patients who underwent double valve replacement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with a sutureless aortic valve implanted in the Cardiovascular and Thoracic Surgery Department of Dijon CHU
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
presence of conduction disorders on postoperative ECGs | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bouchot O, Petrosyan A, Morgant MC, Malapert G. Technical points for aortic valve replacement through right anterior minithoracotomy. Eur J Cardiothorac Surg. 2018 May 1;53(suppl_2):ii24-ii26. doi: 10.1093/ejcts/ezy105. PMID 29718234